CLINICAL TRIAL: NCT07235241
Title: The Effect of Digital Game-Based Teaching Methods on the Development of Ethical Sensitivity and Ethical Decision-Making Processes in Nursing Students
Brief Title: The Effect of Digital Games on Ethical Sensitivity and Decision Making in Nursing Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Furkan Keles, MSc, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IMU17
Record Dates: First submitted 2025-11-13; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Decision Making; Ethics
Keywords: Ethics; Decision Making; Digital Game; Nursing Students

STUDY DESIGN:
Intervention Model Description: A total of two groups, comprising one experimental group and one control group
Who Masked: Participant
Masking Description: Participants do not know which group they will be in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Both the experimental and comparison groups will receive a reminder lecture from the researcher on ethical principles and codes prior to the applications. Participants in the experimental group will simultaneously play digital games and participate in classroom group work after the reminder lesson.
  Interventions: Other: Digital game; Other: In-class group work
- Comparison (Other): They will only participate in in-class group work.
  Interventions: Other: In-class group work

INTERVENTIONS:
Other: Digital game — Digital Game:
  The developed digital game aims to enhance medical students' ethical awareness and decision-making skills. The digital game first provides students with reminders about ethical principles.
  The game covers a four-week process, focusing on a specific ethical principle each week. Each weekly module presents two cases supported by animated visuals written by the researcher, reviewed by experts, and created by the software company. After watching and reading the cases, students answer related questions.
  The modules and principles covered are as follows:
  Week 1 (Do No Harm/Beneficence): Cases related to treatment refusal and palliative care compliance.
  Week 2 (Autonomy/Respect): Cases related to organ donation decisions and chemotherapy refusal.
  Week 3 (Justice/Equity): Cases related to resource (air mattress) allocation and patient prioritisation.
  Week 4 (Confidentiality/Privacy): Cases related to HIV diagnosis confidentiality and psychiatric service confidentiality.
  Arms: Experimental group
Other: In-class group work — Face-to-face case analysis will be conducted over 4 weeks. These sessions are scheduled outside the course programme, once a week for 40 minutes.
  A total of 4 cases, each relating to an ethical principle, will be given to students in printed form at the beginning of each session, and they will be asked to analyse them simultaneously. Before the exercises, students will be explained how to analyse the cases.

SUMMARY:
The study was planned using a randomised controlled experimental design to determine the effectiveness of digital game-based teaching in the development of ethical sensitivity and ethical decision-making processes among nursing students.

DETAILED DESCRIPTION:
The most significant contribution this study will make to the literature is its systematic demonstration of the effects of a digital game-based teaching method on the development of ethical sensitivity and ethical decision-making processes in the context of nursing education. Currently, ethics education is mostly conducted using traditional methods, and it is known that students experience difficulties in transferring what they learn in theoretical education to practice. This study makes a unique contribution by demonstrating that digital games can support students' ethical thinking and decision-making skills by offering interactive and experience-based learning opportunities. Furthermore, the study aims to expand the limited literature on the use of digital game-based teaching in ethics education in nursing and to provide evidence-based data on the integration of technological innovations in ethics education. In this respect, the research is of a nature that will strengthen the pedagogical foundations of nursing education and pioneer the development of student-centred and innovative teaching strategies.

ELIGIBILITY:
Inclusion Criteria:

Students must:

* Have taken and successfully completed the Nursing Ethics course,
* Be a fourth-year nursing student who has successfully completed all professional courses and is undertaking the 'Professional Training in the Workplace' placement.

Exclusion Criteria:

* Students who have not taken the Nursing Ethics course or have failed the course before taking the Professional Training in the Workplace course.
* Having a conditional grade point average (CGPA <2.00) up to the period when the data was collected.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Adapted Ethical Sensitivity Scale for Nursing Students | 3 times; a week before implementation, a week after implementation, 2 months after implementation
  This scale determines the ethical sensitivity levels of nursing students.
  The 7-point Likert-type scale (1=Strongly disagree, 7=Strongly agree) consists of 30 items and six subscales. Items 8, 24, and 29 are reverse-scored. The total score ranges from 30 to 210; a high score indicates high ethical sensitivity.
  Item averages are evaluated as 7-5.9 (very important), 5.8-5 (important), 4.9-3.1 (neutral), and below 3.1 (unimportant).
The Ethical Dilemma Test in Nursing | 3 times; a week before implementation, a week after implementation, 2 months after implementation
  The scale developed under the name 'Nursing Dilemma Test' aims to identify ethical issues in nursing and consists of six scenarios.
  Each scenario has three sections (A, B, C):
  Section A (Action): Measures the decision to be made in the face of an ethical dilemma (to act/not to act/to be undecided).
  Section B (Thinking Style): Determines the 'Principled Thinking' (NPT - importance given to ethical principles) and 'Practical Thinking' (PT - importance given to environmental factors) scores by ranking six statements based on Kohlberg's theory.
  Section C (Familiarity): Calculates the 'familiarity' score by questioning the case experience.
  Scoring:
  NPT Score: ranges from 18 to 66. PT Score: ranges from 6 to 36. Familiarity Score: 6-17 (familiar), 18-30 (unfamiliar).
  Reliability (Turkish Version):
  Cronbach's Alpha: NPT (0.59), PT (0.50). Test-Retest: NPT (0.77), PT (0.73).

SECONDARY OUTCOMES:
Student Satisfaction and Self-Confidence in Learning Scale | Once; a week after implementation
  This scale assesses students' satisfaction with education and their attitudes towards self-confidence in learning.
  The 5-point Likert-type scale (1=Strongly disagree, 5=Strongly agree), consisting of 13 items in total, has two subscales:
  Satisfaction with Learning (5 items) Self-Confidence (8 items)
  Items are reverse-coded. The total score ranges from 13 to 65; a high score indicates high satisfaction and self-confidence. The Cronbach's alpha coefficients of the original scale were found to be Satisfaction (0.94) and Self-Confidence (0.87).
  The Cronbach's alpha values for the Turkish form were found to be Satisfaction (0.89), Self-Confidence (0.83), and Scale Total (0.90).

CONTACTS AND LOCATIONS:
Overall Officials: Furkan Keles, PhD Student, Principal Investigator — Istanbul University - Cerrahpasa; Funda Büyükyılmaz, Prof. Dr., Principal Investigator — Istanbul University - Cerrahpasa

IPD SHARING:
Plan to Share IPD: No